CLINICAL TRIAL: NCT06964542
Title: Effect of Supervised in Comparison to Non-supervised Multicomponent Exercise Training on Balance and Quality of Life in Peripheral Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/63
Record Dates: First submitted 2025-05-01; First posted 2025-05-09 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Peripheral Diabetic Neuropathy
Keywords: Endurance; Multicomponent exercise training; Diabetes Mellitus; Peripheral Diabetic Neuropathy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised Group (Experimental): In supervised exercise intervention a multicomponent exercise training will be applied to group 1 patients for improveent of symptoms caused from diabetic peripheral neuropathy such as balance, endurance, strength and quality of life. Strength and resistive training along with aerobic and balance training will be applied to patients under the supervision of physical therapist in a clinical setup.
  Interventions: Procedure: Multicomponent exercise intervention
- NON SUPERVISED (Experimental): In non-supervised exercise training, patients will receive multicomponent exercise intervention without the supervision of physical therapist but still under the supervision of caregiver at home. Patients will be provided with the complete guidance in the form of exercise diary. This diary included all the protocols for exercise at home , it also included QR code.
  Interventions: Procedure: Non Supervised

INTERVENTIONS:
Procedure: Multicomponent exercise intervention — Patient will be under the complete supervision of physical therapist in a clinical setup.A total of 18 sessions of supervised multicomponent exercise training, thrice a week on alternate days for 6 consecutive weeks, session will be of 45 mins. Multicomponent exercise training including strength and progressive resistance training exercises, actvities will inc. Seated Marching,heel raises,toe raises, sit - to-stand. And balance training activities will involve tandem stands,single leg stance,weight shifting and resistance activities including weight lifting according to feasibility.
  Arms: Supervised Group
Procedure: Non Supervised — In non supervised group , patient will receive all the intervention with the help of exercise diary and guidance provided by the physical therapist. Patient will perform 18 sessions, thrice a week on alternative days, for 6 consecutive days for 45 mins. In diary patient is provided the tick mark table in which patient will mark the attendance on days ptn will perform the exercise. Diary is a complete guidance for home based exercise program which include QR based videos of performance of all exercises and complete guidelines are provided in urdu for the better understanding along with pictorial information. In this program activities that patient will perform includes; stairs climbing, sit to stand, leg raises, side stepping, leg raises with weight on ankles starting from 1kg to 3kg. Walk starting from 20 minutes to 40 minutes till 6 weeks. Resistance and other activities will be included.
  Arms: NON SUPERVISED

SUMMARY:
THIS STUDY IS A RANDOMIZED CONTROL TRIAL AND THE PURPOSE OF THIS STUDY IS TO DETERMINE THE effect of supervised in comparison to non-supervised multicomponent exercise training on balance and quality of life in peripheral diabetic neuropathy

DETAILED DESCRIPTION:
Effect of exercises to assess the benefits on strength endurance, balance and mobility.

Peripheral Neuropathy aged 55-70 will be recruited in the study. The participants would be assessed through WHOQOL BREF, BERG BALANCE SCALE, TIME UP AND GO TEST .

Informed Consent will Be taken after which the participants will be recruited into the two groups, where one group will receive supervised exercise intervention while other group will receive non supervised exercise intervention

ELIGIBILITY:
Inclusion Criteria:

* Age 55-70 years (both male and female)
* Diagnosed patients of diabetes type 2, 10 years after disease
* Completely assessed with Michigan Neuropathy Screening Instrument (MNSI) score scale and patients fulfilling this criterion will be included in this study
* Patients who are fulfilling PARQ will be included in study

Exclusion Criteria:

* Hypoglycemia
* Patient having ischemic heart diseases will not be included
* unable to walk independent
* major orthopedic problems (e.g. lower limb fractures)
* Diagnosed neurological and psychological patients

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Balance | 4 weeks
  Berg balance scale. The score range is 0-56, with higher scores indicating better balance and functional mobility.
Strength | 4 weeks
  The MMT scale refers to the Manual Muscle Testing scale, a standardized method used by physical therapists and healthcare providers to assess muscle strength. It has 6 grades.
ENDURANCE | 4 weeks
  6-Minute Walk Test (6MWT) ) is a widely used and validated test to assess endurance.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Thrapy, Islamabad, Pakistan